CLINICAL TRIAL: NCT04112875
Title: Effect of L-arginine Supplementation on Microcirculation, Endothelial Function and Vascular Smooth Muscle of Young, Elderly and Patients With Sarcopenia and Type 2 Diabetes Mellitus
Brief Title: Effect of L-arginine on Microcirculation, Myogenesis and Angiogenesis Associated With Aging, Sarcopenia and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Laboratory for Clinical and Experimental Research on Vascular Biology (Unknown)
Responsible Party: Principal Investigator, Gerusa Maritimo da Costa, Principal Investigator, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Arginine
Record Dates: First submitted 2019-09-25; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Aging; Sarcopenia; Type 2 Diabetes; Microcirculation
Keywords: L-arginine; Asymmetric Dimethylarginine; Arginase; Sarcopenia; Myostatin; Follistatin; Type 2 diabetes mellitus; Vascular smooth muscle; endothelial function
MeSH Terms: conditions — Sarcopenia; Diabetes Mellitus, Type 2 | interventions — Arginine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-arginine (Active Comparator): L-arginine supplementation: 5g/sachet with water 30 minutes before breakfast for 14 days.
  Interventions: Dietary Supplement: L-arginine
- Maltodextrin (Placebo Comparator): Maltodextrin supplementation: 5g/sachet with water 30 minutes before breakfast for 14 days.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: L-arginine — Handled powdered supplement to be mixed with water, has orange flavor for oral use.
  Arms: L-arginine
Dietary Supplement: Maltodextrin — hydrolysis of cornstarch or starch as a white powder to be mixed with water, has orange flavor for oral use.
  Arms: Maltodextrin

SUMMARY:
This study aims was evaluated the effect of L-arginine on microcirculation, vasoreactivity / endothelial function and vascular smooth muscle of young and old women with Sarcopenia or Type 2 Diabetes Mellitus measured by Nailfold videocapillaroscopy and venous occlusion plethysmography before and after 14 days of consumption 5g oral L-arginine supplementation.

DETAILED DESCRIPTION:
Aging causes responsible endothelial changes, in part by a decrease in the blood flow of the skeletal muscles of the elderly. Reduction of muscle mass / function (Sarcopenia) and Diabetes Mellitus are frequent pathologies in the elderly. L-Arginine is a semi-essential amino acid precursor to nitric oxide synthesis (NO), an important vasodilator and protector cardiovascular.

Seventy-five women were allocated into three groups: twenty-five healthy young (HY) recruited among University students, and fifty women elderly, this was stratified in twenty-five healthy elderly (HE) control and twenty-five with hyperglycemia (HG) elderly from the ambulatories of the Geriatric and Diabetology at the State University of Rio de Janeiro (UERJ) and private supplementary health program. To control group was considered absence cardiovascular risk factor except advanced age. Participants were subjected to screening phase before being eligible for the study by telephone, which comprised of individual clinical history. All subjects signed the written Informed Consent Form enclosed in the protocol approved by Ethics Committee from the State University of Rio de Janeiro according to Helsinki Declaration.

The subjects elected for research made 4 visits to the Biovasc laboratory for data collection. First day: the protocol was explained and agreement from the voluntary obtained, followed and anamnesis and physical exam that included measure at-rest blood pressure, weight and height. Moreover, women examined after 6 hours fasting the microcirculation function using nailfold vidiocapilaroscopy (NVC), followed of the measure of forearm blood flow (FBF) and vascular reactivity by venous occlusion plethysmography (VOP). Second day: Venous blood sample collection after 12 hours fasting. In sequence, they realized whole-body dual-energy X-ray absorptiometry (DXA) to calculate the body composition main measure lean and fat mass. After, was delivered a box with 14 sachets content 5g L-arginine supplementation, and it was recommended to ingest with water 30 minutes before breakfast during 14 days. Third day: Return after the supplementation to realize measurement weight, and exams NVC and VOP. Fourth day: blood sample were taken after 12 hours fasting under effect of the L-arginine.

ELIGIBILITY:
Inclusion Criteria:

* young women aged between 20 - 30 years, IMC < 24.9 kg/m2
* older women over 65 years healthy, BMI <35 kg/m2.
* Elderly women with or without a preexisting diagnosis of diabetes mellitus with fasting plasma glucose (FPG) > 100 mg/dL were classified into type 2 diabetes mellitus.

Exclusion Criteria:

* involved type 1 diabetes mellitus
* insulin use, cognitive impairment
* frailty
* disorders cardiometabolic
* liver and/or kidney dysfunction
* autoimmune diseases
* smoking
* rigorous exercise
* uncontrolled hypertension with pressure level > 140/90 mmHg, with up to two antihypertensive drugs of different classes.

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Changes in Microcirculation | before and after 14 days of intervention
  Assessing microvascular changes in the peripheral circulation by microcirculatory image recordings were used Nailfold vidiocapilaroscopy.
Changes in Endothelium-dependent and endothelium-independent vasodilation | before and after 14 days of intervention
  Changes in vasodilatation by endothelial reactivity and smooth muscle responsiveness were assessed by Venous occlusion plethysmography

SECONDARY OUTCOMES:
Change in metabolic markers | before and after 14 days of intervention
  Metabolic markers associated with lipid profile (total cholesterol, triglycerides, Low Density Lipoproteins (HDLc) and High Density Lipoproteins (LDLc)); renal profile (urea and creatinine); Glycemic and insulin were analyzed to verify treatment response by comparing the results (mg/dL) before and after oral supplementation in the studied groups.
change in circulating muscle growth and degradation factors | before and after 14 days of intervention
  Insulin-like growth factor-I (IGF-I) and follistatin (Fslt-I) growth-associated and (GDF-8 / Myostatin and interleukin 6 (IL-6)) degradation-associated were analyzed to verify response to treatment, comparing results (ng / ml) before and after oral supplementation in the study groups.
Body composition by DXA | before of intervention
  The whole-body dual-energy X-ray absorptiometry (DXA) was used to measure appendicular skeletal muscle (ASM) composed lean body mass of arms and legs to calculated skeletal muscle mass index by following formula: ASM/height2.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Bottino, PhD, Principal Investigator — State University of Rio de Janeiro; Gerusa M Costa, MSc, Principal Investigator — State University of Rio de Janeiro
Locations (1):
- State University of Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.